CLINICAL TRIAL: NCT05290740
Title: Comparison of Two Norepinephrine Rescue Bolus Doses for Management of Severe Post-spinal Hypotension During Elective Cesarean Delivery: A Randomized, Controlled Trial
Brief Title: Two Norepinephrine Rescue Bolus Doses for Management of Severe Post-spinal Hypotension During Elective Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-657-2021
Record Dates: First submitted 2022-02-22; First posted 2022-03-22 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Postspinal Hypotension; Cesarean Delivery; Norepinephrine
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator)
  Interventions: Drug: Norepinephrine 5 mcg
- group B (Active Comparator)
  Interventions: Drug: Norepinephrine 10 mcg

INTERVENTIONS:
Drug: Norepinephrine 5 mcg — norepinephrine bolus of 5 mcg for treatment of sever postspinal hypotension
  Arms: group A
Drug: Norepinephrine 10 mcg — norepinephrine bolus of 10 mcg for treatment of sever postspinal hypotension
  Arms: group B

SUMMARY:
Maternal hypotension after spinal block is a common complication after subarachnoid block in this population whose incidence reached 60% in many reports. Hypotension is associated with maternal and neonatal complications; therefore, it is highly recommended to use vasopressors, prophylactically and interactively, for prompt control maternal blood pressure. Despite the presence of various preventive regimens (fluid loading, maternal positioning, and vasopressors), many mothers develop intraoperative episodes of hypotension which requires the use of a vasopressor bolus.

Norepinephrine (NE) is an alpha adrenergic agonist with weak beta adrenergic agonistic activity; and is increasingly used in obstetric anesthesia with acceptable maternal and neonatal outcomes. NE bolus could be used for rapid correction of maternal blood pressure in a dose which variedranged between 3.7-10 mcg. Till date, al the available data for the management of maternal hypotension did not differentiate between severe and non-severe hypotension. The incidence of severe maternal hypotension (systolic blood pressure ≤60% of baseline) ranged between 7-20%. In a recent report, Hassabelnaby et al compared 6 mcg and 10 mcg NE boluses in management of maternal hypotension and found that the doses had the same success rate (≈90%); however, most of the participants in the mentioned study had non-severe hypotension. Therefore, we hypothesize that severe hypotension should be separately investigated for the possible superiority of the higher over the lower dose of NE bolus.

Insufficient NE bolus would lead to failed management and prolonged hypotensive episode, whereas a higher dose might lead to reactive hypertension and/or bradycardia, which is sometimes severe. Therefore, determining the optimum dose for NE bolus would enable proper control of maternal hemodynamic profile

DETAILED DESCRIPTION:
Upon arrival to the operating room, the patient will be in supine position with left uterine displacement using a wedge below the right buttock. Routine monitoring will be applied (electrocardiography, pulse oximetry, and non-invasive blood pressure monitor). An 18G-cannula will be inserted, and the patients will receive 10 mg metoclopramide. Baseline heart rate and systolic blood pressure will be recorded as the average of three consecutive readings with 2-minutes interval.

Lactated Ringer's solution will be infused at rate of 15 mL/Kg over 10 minutes as a co-load; spinal anesthesia will be achieved by injecting 10 mg of hyperbaric bupivacaine and 20 mcg fentanyl into the subarachnoid space at L3-L4 or L4-L5 interspace using 25G spinal needle.

After subarachnoid block, mothers will be placed in the supine position with left-lateral tilt. The decision to give prophylactic vasopressor infusion will be according to the attending anesthetist preferences.

Block success will be assessed after 5 minutes from intrathecal injection of local anesthetic; and will be confirmed if sensory block level is at T4.

The patient would receive the study drug only if she developed severe post-spinal hypotension (defined as systolic blood pressure ≤60% of the baseline reading) as her first hypotensive episode or after 10 minutes from the last successfully managed hypotensive episode and before the delivery. .

The management of the hypotensive episode will be considered successful if the systolic blood pressure is > 80% of the baseline within 2 mins of the bolus. If the bolus failed, NE bolus of 5 mcg will be given.

Any other hypotensive episode (systolic blood pressure <80% of baseline) will be managed with NE bolus of 5 mcg.

Intraoperative bradycardia (defined as heart rate less than 55 bpm) will be managed by IV atropine bolus (0.5 mg) will be administered.

Fluid administration will be continued up to a maximum of 1.5 liters. An oxytocin bolus (0.5 IU) will be delivered over five seconds after delivery then infused at a rate of 2.5 IU/hour.

ELIGIBILITY:
Inclusion Criteria:

* full-term singleton pregnant women
* American society of anesthesiologist physical status of I or II,
* scheduled for elective cesarean delivery

Exclusion Criteria:

* Patients with uncontrolled cardiac morbidities (patients with tight valvular lesion, impaired contractility with ejection fraction < 50%, heart block, and arrhythmias),
* hypertensive disorders of pregnancy,
* peripartum bleeding, coagulation disorders (patients with INR >1.4 and or platelet count < 80000 /dL) or
* any contraindication to regional anesthesia, and
* baseline systolic blood pressure (SBP) < 100 mmHg

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
incidence of successful management of severe post-spinal hypotension | 2 minutes after drug injection
  systolic blood pressure >80% of baseline within 2 min of drug injection

SECONDARY OUTCOMES:
time to severe postspinal hypotension | 1 minute after subarachnoid local anesthetic injection till 1 min after baby delivery
  minutes
incidence of reactive bradycardia | 2 minutes after drug injection
  heart rate heart rate less than 55 beat per minute
incidence of reactive hypertension | 2 minutes after drug injection
  systolic blood pressure >120% of baseline
incidence of nausea and vomiting | 1 minute after subarachnoid local anesthetic injection till 5 minute after baby delivery
  unpleasant painless subjective feeling that one will imminently vomit or vomiting
fetal umbilical blood pH | at 5 minutes post delivery
  pH
baby Apgar score | at 5 minutes post delivery
  score with 0, 1, or 2, depending on the observed condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
protocol and data of this research could be available from the PI upon reasonable request

REFERENCES:
- [Derived] Amin SM, Hasanin A, Ghanem NT, Mostafa M, Elzayat N, Elsherbiny M, Abdelwahab Y. Comparison of Two Norepinephrine Rescue Bolus Doses for Management of Severe Post-Spinal Hypotension During Elective Caesarean Delivery: A Randomized, Controlled Trial. Int J Gen Med. 2024 Jan 19;17:153-160. doi: 10.2147/IJGM.S446021. eCollection 2024. PMID 38264276